CLINICAL TRIAL: NCT00403559
Title: A 4 Week Randomized Double-blind Parallel Group Active Comparator Controlled Study of Elidel (Pimecrolimus) for the Treatment of Seborrheic Dermatitis
Brief Title: A 4 Week Study of Elidel (Pimecrolimus) for the Treatment of Seborrheic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermatology Specialists Research (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CUS37; SAIRB # 06-4893 (Other: DematologySR); IND 75,225 (Other: DematologySR)
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Seborrheic Dermatitis
Keywords: seborrheic dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic | interventions — pimecrolimus; Ketoconazole

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elidel Cream (pimecrolimus) (Experimental): Elidel Cream to be applied twice daily for 4 weeks
  Interventions: Drug: Elidel
- Ketoconazole Cream (Nizoral) (Active Comparator): Ketoconazole Cream to be applied twice daily for 4 weeks
  Interventions: Drug: Ketoconazole Cream

INTERVENTIONS:
Drug: Elidel
  Other Names: pimecrolimus
  Arms: Elidel Cream (pimecrolimus)
Drug: Ketoconazole Cream
  Other Names: Nizoral
  Arms: Ketoconazole Cream (Nizoral)

SUMMARY:
This is an exploratory study to determine effectiveness of Elidel for the treatment of seborrheic dermatitis

DETAILED DESCRIPTION:
This is a 4 week study for patients 18 and older to compare the efficacy and safety of pimecrolimus cream 1% twice daily and ketaconazole cream 2 % twice daily for the treatment of seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 or older and sign written informed consent.
* Must be wiling and able to comply with protocol.
* Must have active seborrheic dermatitis of the face.

Exclusion Criteria:

* No history of overt bacterial, viral or fungal infection of the head/neck.
* No history or presence of compromising dermatosis elsewhere on the skin
* No Parkinson's disease, HIV, infections or disorders of the central nervous system
* No actinically damaged skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-05-07 (Actual); Primary Completion 2009-02-20 (Actual); Study Completion 2009-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kempers, MD, Principal Investigator — Associated Skin Care Specialists; Bernard Goffe, MD, Principal Investigator — Dermatology Associates; Debra Breneman, MD, Principal Investigator — University of Cincinnati - Dermatology
Locations (1):
- Dermatology Specialists, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began in May 2007. All subject visits were completed by Feb. 2009. There were 4 research sites, all part of dermatology practices. Subjects were recruited from the patient population of each site.
Pre-assignment Details: Consented subjects who had been using topical medication for their seborrheic dermatitis, underwent withdrawal from this treatment (washout) for 2 weeks prior to being randomized and beginning use of study product. One subject after undergoing washout did not qualify for randomization due to not meeting disease severity criteria. This subject was not included in the total number of subjects who started the study.
Groups:
- Elidel Cream: Participants randomly assigned Elidel Cream twice daily for four weeks.
- Ketoconazole Cream: Participants randomly selected to apply Ketoconazole Cream twice daily for 4 weeks.
Period: Overall Study
Arm/Group | Elidel Cream | Ketoconazole Cream
Started | 56 | 56
Completed | 52 | 52
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Elidel Cream 1%: In a randomized fashion, fifty six participants with facial seborrheic dermatitis were assigned to Elidel Cream 1% (pimecrolimus) to be applied twice daily for 4 weeks
- Ketoconazole Cream 2%: n a randomized fashion, fifty six participants with facial seborrheic dermatitis were assigned to Ketoconazole Cream 2% to be applied twice daily for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Elidel Cream 1% | Ketoconazole Cream 2% | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 11 | 11 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 27
  Male | 39 | 46 | 85
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 112

OUTCOME MEASURES:

1. Primary Outcome: The Change of F-IGA From Baseline (BL) to wk 1 Will be the Primary Efficacy Variable.
Description: F-IGA is defined as Facial Investigator's Global Assessment, which incorporates assessments of the severity of facial seborrheic dermatitis. Scoring is 0 to 3, 0 describing a better outcome with progressively worsening up to 3 representing a worse outcome (whole number only). 0 = Clear; 1 = Mild; 2 = Moderate and 3 = Severe. Scoring is based upon morphologic description of signs of erythema (0 =none, 1= faint, 2 =dull, 3 =deep/dark red) and scaling (0 = none, 1 = minute, powdery scale, 2 = thin flakes of scale, 3 = scales covering most of the involved areas).
Time Frame: One week from Baseline
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Elidel (Pimecrolimus) Cream 1% Arm: The Change in F-IGA from BL to Wk 1 assigned Elidel Cream (pimecrolimus) 1%
- Ketoconazole Cream 2% Arm: The Change in F-IGA from BL to Wk 1 assigned Ketoconazole Cream 2%
Arm/Group | Elidel (Pimecrolimus) Cream 1% Arm | Ketoconazole Cream 2% Arm
Number analyzed (Participants) | 56 | 56
units on a scale | -0.9 (0.8) | -0.6 (0.7)
Statistical Analysis 1: Comparison: Elidel (Pimecrolimus) Cream 1% Arm vs Ketoconazole Cream 2% Arm; Test type: Non-Inferiority — Non-inferiority determined as the F-IGA, IGA, erythema, scaling, and pruritis scores when compared between groups. The Wilcoxon rank sum test stratified baseline seborrheic dermatitis (SD) severity; p = .009, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Key Secondary Efficacy Will be the % of Patients With Facial Clearance
Description: Number of participants in each arm (Elidel vs Ketoconazole) who achieved total facial clearance.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Elidel Cream (Pimecrolimus): Elidel Cream to be applied twice daily for 4 weeks
  Elidel
- Ketoconazole Cream (Nizoral): Ketoconazole Cream to be applied twice daily for 4 weeks
  Ketoconazole Cream
Arm/Group | Elidel Cream (Pimecrolimus) | Ketoconazole Cream (Nizoral)
Number analyzed (Participants) | 56 | 56
participants | 56 | 56

ADVERSE EVENTS:
Time Frame: 4 weeks per subject, Baseline to End of Study
Description: Definitions as per www.ClinicalTrials.gov
Groups:
- Elidel Cream: Elidel (pimecrolimus) Cream 1% Arm
- Ketoconazole Cream: Ketoconazole Cream 2% Arm
Arm/Group | Elidel Cream | Ketoconazole Cream
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 16/56 | 9/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elidel Cream (N=56) | Ketoconazole Cream (N=56)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Facial redness
Facial skin flaking (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Area of study medication application
Burning sensation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Immediate burning sensation upon application of study medication, resolves within 15 minutes
Feeling of warmth (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — Site application had a sensation of warmth
Dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Facial skin dry at area of study medication application
Common Cold (Infections and infestations) | 1 (1) | 2 (2) — Symptoms of nasal congestion and excessive drainage during course.
Sore throat (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Fracture of lower extremity bones
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Area of study medication application
Muscular Ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (General disorders) | 0 (0) | 1 (1)
Domestic animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Rectal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash not at study medication application site
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nodular basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1)
Dry Eyes (Eye disorders) | 1 (1) | 0 (0)
Loss of Balance (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Hive on non study medication application site
Pain Left Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Trial limitations: patient usage diaries may not have been accurate. Greater improvement may have been seen in either arm with a longer trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No